CLINICAL TRIAL: NCT00130533
Title: Multicenter, Open-label, Randomized Phase III to Evaluate Efficacy of Maintenance Treatment With Capecitabine Following Standard Adjuvant Chemotherapy in Operable Triple Negative Breast Cancer Patients
Brief Title: Maintenance Treatment With Capecitabine Versus Observation in Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Hoffmann-La Roche (Industry); IBEROAMERICAN COALITION FOR BREAST ONCOLOGY RESEARCH (CIBOMA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBOMA 2004-01; 2005-002838-36 (EudraCT Number)
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Triple-Negative Early Breast Cancer; Maintenance Adjuvant Chemotherapy; Capecitabine; Basal-like genotype; Triple-Negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

ARMS (2):
- Xeloda (capecitabine) (Experimental): 1000 mgrs/m2 twice a day, tablets, 8 cycles
  Interventions: Drug: Capecitabine
- Observation (No Intervention): Observation. No intervention.

INTERVENTIONS:
Drug: Capecitabine
  Other Names: Xeloda
  Arms: Xeloda (capecitabine)

SUMMARY:
This is a prospective, open-label, randomized phase III study assessing adjuvant capecitabine after standard chemotherapy for patients with early triple negative breast cancer.

DETAILED DESCRIPTION:
Patients will be stratified as per investigational site, previous adjuvant chemotherapy (anthracyclines versus anthracyclines plus taxanes), and number of affected axillary lymph nodes (0, 1-3, >= 4). Node negative patients must present a tumour size > 2 cm to be eligible. At least 6 lymph nodes must be analysed to confirm the number of affected nodes. Patients will be randomised to receive: 8 courses of capecitabine 1000 mg/m2 by mouth, twice a day (p.o. bid) for 14 days, followed by a 7 day rest versus observation.

Tissue samples must be analysed by a central laboratory, to confirm estrogen receptor (ER), progesterone receptor (PgR), human epidermal growth factor receptor-2 (HER2), cytokeratins (CK) 5/6 and epidermal growth factor receptor (EGFR) status.

The following data were obtained from the database of the "El Alamo" project. One thousand six hundred and twenty-seven (1,627) in total were considered during the years 1990 to 1997. The population is formed of patients with operable breast cancer, with surgery, positive nodes, and negative hormone receptors, or negative nodes, negative hormone receptors and T2-3 tumors.

For these patient groups, estimated 5-year disease-free survival is 64.72%. Assuming an exponential distribution, the aim is to detect an increase of 64.72% to 73.7% in 5 years Disease Free survival rate corresponds to a Hazard Ratio of 0.701 and a risk reduction of about 30%, with a power of 80% using a two-tailed log-rank test at 0.05 and whereas 4 years of recruitment period and 3 years of follow-up period. We would need 255 events, 834 patients without considering any dropouts.

Considering a drop-out rate of 5% post-randomization, the final sample size will be 876 patients, 438 per treatment arm.

The sample size calculation was performed by the program package "EAST" version 5.2.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Histological diagnoses of operable invasive adenocarcinoma of the breast (T1-T3). Tumours must be HER2 negative. Time window between end of adjuvant chemotherapy and study randomization must be less than 8 weeks. In patients receiving adjuvant radiotherapy, time window allowed between last session and randomisation is 4 weeks.
* Surgery must consist of mastectomy or conservative surgery with axillary lymph node dissection. Margins free of disease and ductal carcinoma in-situ (DCIS) are required. Lobular carcinoma is not considered a positive margin.
* Node negative patients with tumour size > 2 cm.
* Positive axillary lymph nodes defined as at least 1 out of 6 nodes with presence of disease. If sentinel node technique is used, sentinel node can be the only node affected. Patients belonging to the following classifications are eligible: pN1a (Metastases in 1-3 axillary lymph nodes, at least one metastasis greater than 2.0 mm), pN2a (Metastases in 4-9 axillary lymph nodes (at least one tumor deposit greater than 2 mm)), pN3a (Metastases in 10 or more axillary lymph nodes [at least one tumor deposit greater than 2 mm]; or metastases to the infraclavicular [level III axillary lymph] nodes).
* Status of hormone receptors in primary tumour. Negative results must be available before the end of adjuvant chemotherapy.
* Patients must not present evidence of metastatic disease.
* Negative status of HER2 in primary tumour, known before randomization.
* Adjuvant chemotherapy consisting of a minimum of 6 courses with anthracyclines and/or taxanes.
* Age >= 18 and <= 70 years old.
* Performance status (Karnofsky index) >= 80.
* Laboratory results (within 14 days prior to randomization):
* Hematology:

  * neutrophils >= 1.5 x 10e9/l;
  * platelets >= 100x 10e9/l;
  * hemoglobin >= 10 mg/dl
* Hepatic function:

  * total bilirubin <= 1 upper normal limit (UNL);
  * Aspartate aminotransferase (AST or SGOT) and Alanine aminotransferase (ALT or SGPT) <= 2.5 UNL;
  * alkaline phosphatase <= 2.5 UNL.
  * If values of SGOT and SGPT > 1.5 UNL are associated to alkaline phosphatase > 2.5 UNL, patient is not eligible.
* Renal Function:

  * creatinine <= 175 µmol/l (2 mg/dl).
  * creatinine clearance >= 60 ml/min.
* Pharmacogenetics:

  * one blood sample is needed for single nucleotide polymorphism (SNP) assessment.
* Patients able to comply with treatment and study follow-up.
* Negative pregnancy test done in the 14 previous days to randomization.

Exclusion Criteria:

* Prior therapy with anthracyclines or taxanes (paclitaxel or docetaxel) for any malignancy.
* Pregnant or lactating women. Adequate contraceptive methods must be used during chemotherapy and hormone therapy treatments. Negative pregnancy test in the 14 previous days to randomization.
* Bilateral invasive breast cancer.
* Any T4 or M1 tumour.
* Axillary lymph nodes: patients belonging to the following classifications are excluded: pN1b (Metastases in internal mammary nodes with micrometastases or macrometastases detected by sentinel lymph node biopsy but not clinically detected), pN1c (Metastases in 1-3 axillary lymph nodes and in internal mammary lymph nodes with micrometastases or macrometastases detected by sentinel lymph node biopsy but not clinically detected), pN2b (Metastases in clinically detected internal mammary lymph nodes in the absence of axillary lymph node metastases), pN3b (Metastases in clinically detected ipsilateral internal mammary lymph nodes in the presence of one or more positive axillary lymph nodes; or in more than three axillary lymph nodes and in internal mammary lymph nodes with micrometastases or macrometastases detected by sentinel lymph node biopsy but not clinically detected), pN3c (Metastases in ipsilateral supraclavicular lymph nodes).
* Any other serious medical pathology, such as congestive heart failure, unstable angina, history of myocardial infarction during the previous year, uncontrolled hypertension or high risk arrhythmias.
* History of neurological or psychiatric disorders, which could preclude the patients to free informed consent.
* Active uncontrolled infection.
* Active peptic ulcer, unstable diabetes mellitus.
* Previous or current history of neoplasms different to breast cancer, except for skin carcinoma, cervical in situ carcinoma, or any other tumour curatively treated and without recurrence in the last 10 years; ductal in situ carcinoma in the same breast; lobular in situ carcinoma.
* History of hypersensitivity to capecitabine, fluorouracil.
* Patients lacking physical integrity of upper gastrointestinal tract or with history of bad absorption syndrome.
* History of dihydropyrimidine dehydrogenase (DPD) deficiency.
* Anticoagulant treatment with coumadin anticoagulants.
* Current treatment with sorivudine or its chemical family.
* Concomitant treatment with other investigational products. Participation in other clinical trials with a non-marketed drug in the 30 previous days before randomization.
* Concomitant treatment with other therapy for cancer.
* Males.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Principal Investigator, Principal Investigator — Hospital Clínico Universitario de Valencia
Locations (48):
- Spain (48):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Instituto Catalán de Oncología de L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital del Espíritu Santo, Santa Coloma de Gramenet, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital General de Jerez, Jerez de la Frontera, Cádiz
  - Onkologikoa, Donostia / San Sebastian, Guipúzcoa
  - Hospital de Donostia, Donostia / San Sebastian, Guipúzcoa
  - Hospital de Barbastro, Barbastro, Huesca
  - Hospital Insular de Las Palmas de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Coalición Iberoamericana de Investigación en Oncología Mamaria (CIBOMA), San Sebastián de los Reyes, Madrid
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Oncológico de Galicia, A Coruña
  - Hospital Universitario General de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital Universitario General Yagüe, Burgos
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital de Madrid Norte Sanchinarro (CIOCC), Madrid
  - Hospital Universitario Virgen de la Arrixaca, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Hospitalario de Ourense, Ourense
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario de Valme, Seville
  - Hospital Virgen de la Salud, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Provincial de Zamora "Rodríguez Chamorro", Zamora
  - Hospital Clínico Universitario de Zaragoza "Lozano Blesa", Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Result] Lluch A, Barrios CH, Torrecillas L, Ruiz-Borrego M, Bines J, Segalla J, Guerrero-Zotano A, Garcia-Saenz JA, Torres R, de la Haba J, Garcia-Martinez E, Gomez HL, Llombart A, Bofill JS, Baena-Canada JM, Barnadas A, Calvo L, Perez-Michel L, Ramos M, Fernandez I, Rodriguez-Lescure A, Cardenas J, Vinholes J, Martinez de Duenas E, Godes MJ, Segui MA, Anton A, Lopez-Alvarez P, Moncayo J, Amorim G, Villar E, Reyes S, Sampaio C, Cardemil B, Escudero MJ, Bezares S, Carrasco E, Martin M; GEICAM Spanish Breast Cancer Group; CIBOMA (Iberoamerican Coalition for Research in Breast Oncology); LACOG (Latin American Cooperative Oncology Group). Phase III Trial of Adjuvant Capecitabine After Standard Neo-/Adjuvant Chemotherapy in Patients With Early Triple-Negative Breast Cancer (GEICAM/2003-11_CIBOMA/2004-01). J Clin Oncol. 2020 Jan 20;38(3):203-213. doi: 10.1200/JCO.19.00904. Epub 2019 Dec 5. PMID 31804894
- [Result] Schettini F, Chic N, Braso-Maristany F, Pare L, Pascual T, Conte B, Martinez-Saez O, Adamo B, Vidal M, Barnadas E, Fernandez-Martinez A, Gonzalez-Farre B, Sanfeliu E, Cejalvo JM, Perrone G, Sabarese G, Zalfa F, Peg V, Fasani R, Villagrasa P, Gavila J, Barrios CH, Lluch A, Martin M, Locci M, De Placido S, Prat A. Clinical, pathological, and PAM50 gene expression features of HER2-low breast cancer. NPJ Breast Cancer. 2021 Jan 4;7(1):1. doi: 10.1038/s41523-020-00208-2. PMID 33397968
- [Result] Asleh K, Lluch A, Goytain A, Barrios C, Wang XQ, Torrecillas L, Gao D, Ruiz-Borrego M, Leung S, Bines J, Guerrero-Zotano A, Garcia-Saenz JA, Cejalvo JM, Herranz J, Torres R, Haba-Rodriguez J, Ayala F, Gomez H, Rojo F, Nielsen TO, Martin M. Triple-Negative PAM50 Non-Basal Breast Cancer Subtype Predicts Benefit from Extended Adjuvant Capecitabine. Clin Cancer Res. 2023 Jan 17;29(2):389-400. doi: 10.1158/1078-0432.CCR-22-2191. PMID 36346687
- [Result] Ye F, Bian L, Wen J, Yu P, Li N, Xie X, Wang X. Additional capecitabine use in early-stage triple negative breast cancer patients receiving standard chemotherapy: a new era? A meta-analysis of randomized controlled trials. BMC Cancer. 2022 Mar 12;22(1):261. doi: 10.1186/s12885-022-09326-5. PMID 35279130
- See also: Sponsor's web — http://www.ciboma.org/
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2006 and September 2011, 876 patients were recruited, across 80 institutions in 8 countries (Spain, Brazil, Chile, Colombia, Ecuador, Mexico, Peru, and Venezuela)
Groups:
- Xeloda (Capecitabine): 1000 mgrs/m2 twice a day, tablets, 8 cycles
  Capecitabine
Period: Overall Study
Arm/Group | Xeloda (Capecitabine) | Observation
Started | 448 | 428
Completed | 337 | 398
Not Completed | 111 | 30
Not completed — Withdrawal by Subject | 33 | 6
Not completed — Adverse Event | 34 | 1
Not completed — Disease relapse | 9 | 13
Not completed — Interruption of treatment > 3 weeks | 11 | 0
Not completed — Death | 4 | 2
Not completed — Protocol Violation | 5 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Sponsor´s decision | 2 | 0
Not completed — Second Primary Malignancy | 0 | 1
Not completed — Other | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xeloda (Capecitabine) | Observation | Total
Number analyzed (Participants) | 448 | 428 | 876
Age, Continuous [Median (Full Range); unit: years] | 50 [20 to 79] | 49 [23 to 82] | 49 [20 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 448 | 428 | 876
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 313 | 309 | 622
  Hispanic | 107 | 97 | 204
  Black | 16 | 11 | 27
  Other | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  Spain | 272 | 260 | 532
  Brazil | 71 | 68 | 139
  Mexico | 61 | 52 | 113
  Chile | 19 | 23 | 42
  Peru | 7 | 12 | 19
  Ecuador | 9 | 9 | 18
  Colombia | 6 | 3 | 9
  Venezuela | 3 | 1 | 4
Karnofsky Index Performance Status [Count of Participants; unit: Participants] — Karnofsky Scale allows patients to be classified as to their functional impairment. The lower the Karnofsky score, the worse the survival for most serious illnesses 100: Normal, no complaints 90: Minor signs or disease symptoms 80: Normal activity with effort 70: Care for self. Unable to carry on normal activity 60: Requires occasional assistance 50: Requires considerable assistance and frequent medical care 40: Disabled. Requires special care and assistance 30: Severly disabled 20: Very sick. Active supportive treatment necessary 10: Moribund 0: Dead
  Participants
    80 | 8 | 17 | 25
    90 | 57 | 67 | 124
    100 | 383 | 344 | 727
Menopausal status at diagnosis [Count of Participants; unit: Participants]
  Premenopausal | 136 | 140 | 276
  Postmenopausal | 312 | 288 | 600
Histologic type [Count of Participants; unit: Participants]
  Invasive ductal carcinoma | 395 | 369 | 764
  Invasive lobular carcinoma | 9 | 10 | 19
  Other | 44 | 49 | 93
Histologic grade [Count of Participants; unit: Participants] — Cancer cells are given a Grade (G) when they are removed from the breast and checked under a microscope. The G is based on how much the cancer cells look like normal cells.
  * G1 or well differentiated (score 3, 4, or 5): cells are slower-growing, and look more like normal breast tissue.
  * G2 or moderately differentiated (score 6, 7): cells are growing at a speed of and look like cells somewhere between G1 and 3.
  * G3 or poorly differentiated (score 8, 9): cells look very different from normal and will probably grow and spread faster.
  Participants
    Grade 1 | 15 | 12 | 27
    Grade 2 | 82 | 81 | 163
    Grade 3 | 323 | 299 | 622
    Unknown | 28 | 36 | 64
Phenotype by immunohistochemistry (IHC) [Count of Participants; unit: Participants] — Basal phenotype: Basal-like tumors receive this name because their genetic expression profile is similar to that of a normal basal epithelial cell. These similarities include the absence of expression of the estrogen receptor and other genes related with this and the human epidermal growth factor receptor 2 (HER2) receptor. They also share with the basal epithelial cells overexpression of cytokeratins 5/6 and 17, epidermal growth factor receptor (EGFR) and genes associated with proliferation. p53 mutations in thyrosine are also basal cell characteristics.
  Participants
    Basal | 319 | 309 | 628
    Non-basal | 129 | 119 | 248
Stage at diagnosis [Count of Participants; unit: Participants] — According to American Joint Committee on Cancer (AJCC) 2002:
  * Stage (S) I: tumour <2 centimetres (cm)
  * S II:
  S IIA: cancer spread to movable ipsilateral axillary (MIA) Lymph Nodes (LN). tumor <2 cm and spread to MIA LN tumor >2 cm but >5 cm
  S IIB:
  tumor >2 cm but <5 cm and spread to MIA LN tumor >5 cm
  - S III: S IIIA: cancer spread to ipsilateral axillary LN fixed or matted S IIIB: tumor spread to the chest wall or caused swelling or ulceration of the breast or is diagnosed as inflammatory breast cancer.
  S IIIC: metastases in ipsilateral infraclavicular LN.
  Participants
    Stage I | 62 | 74 | 136
    Stage II | 270 | 271 | 541
    Stage III | 106 | 80 | 186
    Unknown | 10 | 3 | 13
Nodal status [Count of Participants; unit: Participants]
  Negative | 244 | 242 | 486
  1-3 positive nodes | 121 | 124 | 245
  ≥4 positive nodes | 77 | 61 | 138
  Missing data | 6 | 1 | 7
Type of prior Chemotherapy [Count of Participants; unit: Participants]
  Adjuvant (only) | 353 | 352 | 705
  Neoadjuvant (+/- adjuvant) | 89 | 75 | 164
  Missing data | 6 | 1 | 7
Chemotherapy regimens [Count of Participants; unit: Participants]
  Anthracyclines-based | 147 | 138 | 285
  Anthracyclines and taxanes-based | 301 | 290 | 591
Breast surgery [Count of Participants; unit: Participants]
  Conservative | 237 | 242 | 479
  Mastectomy | 205 | 185 | 390
  Missing data | 6 | 1 | 7
Axillary surgery [Count of Participants; unit: Participants] — axillary lymph node dissection (ALND) sentinel lymph node biopsy (SLNB)
  Participants
    sentinel lymph node biopsy (SLNB) | 99 | 122 | 221
    axillary lymph node dissection +/- SLNB | 349 | 306 | 655
Radiation therapy [Count of Participants; unit: Participants]
  Yes | 352 | 346 | 698
  No | 91 | 81 | 172
  Unknown | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS) Events
Description: DFS was measured from the date of randomization assignment in the intent to treat (ITT) population to loco-regional or distant recurrence, second primary malignancy or death date, whichever occurred first.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Xeloda (Capecitabine) | Observation
Number analyzed (Participants) | 448 | 428
Participants | 105 | 120

2. Secondary Outcome: Disease Free Survival (DFS) Events by Phenotype
Description: as for outcome 1
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Xeloda (Capecitabine) | Observation
Number analyzed (Participants) | 105 | 120
Participants
  Basal Phenotype | 84 | 86
  Non basal Phenotype | 21 | 34

3. Secondary Outcome: Overall Survival (OS) Event
Description: OS event is defined as the death from any cause.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Xeloda (Capecitabine) | Observation
Number analyzed (Participants) | 448 | 428
Participants | 71 | 73

4. Secondary Outcome: The Number of Participants Who Experienced Adverse Events (AE)
Description: Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events).
Time Frame: 5 years
Population: The analysis of toxicity was made in all study patients who had received at least 1 treatment cycle, or who had completed the observation period equivalent to 1 cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | Xeloda (Capecitabine) | Observation
Number analyzed (Participants) | 436 | 425
Participants | 416 | 271

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Xeloda (Capecitabine) | Observation
All-Cause Mortality (participants affected / at risk) | 71/448 | 73/428
Serious Adverse Events (participants affected / at risk) | 23/436 | 6/425
Other Adverse Events (participants affected / at risk) | 416/436 | 271/425
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xeloda (Capecitabine) (N=436) | Observation (N=425)
Gastroenteritis and renal insuficience (Gastrointestinal disorders) | 1 | 0
Supraventricular arrhythmia NOS (Cardiac disorders) | 1 | 0 — Grade 2
Diarrhea (Gastrointestinal disorders) | 4 | 0 — Grade 3
Worsening of depressive syndrome (General disorders) | 1 | 0
Thoracic pain grade 2, disnea G-1 (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection with normal ANC ( Urinary) (Infections and infestations) | 1 | 0 — Grade 3
Neutropenia G 3; Leucopenia G2 (Blood and lymphatic system disorders) | 1 | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 2 | 0 — Grade 5
Hand-foot skin reaction (Nervous system disorders) | 1 | 0 — Grade 3
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Right renal colic (Renal and urinary disorders) | 1 | 0 — Grade 2
Positive pregnant test performed (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Mucositis Oral cavity and Pharynx (Gastrointestinal disorders) | 1 | 0 — Grade 3
Heart failure (Cardiac disorders) | 0 | 1 — Grade 2
Thorax and left arm pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Infarction and cardiac arrest (Cardiac disorders) | 0 | 1
Infection with unknown ANC pulmonary/upper respiratory - lung (pneumonia) (Infections and infestations) | 0 | 1 — Grade 5
Thrombosis/thrombus/embolism: venous thrombosis (Vascular disorders) | 1 | 0 — Grade 3
Ischemia cardiac/Infarction (Cardiac disorders) | 1 | 0 — Grade 3
Axillary nodular resection (Surgical and medical procedures) | 1 | 0
Coronary vasospam (Cardiac disorders) | 1 | 0 — Grade 3
Diarrhea grade 2, Vomiting grade 2, Septic shock grade 5 (Gastrointestinal disorders) | 1 | 0
Showed lumbar column fracture(L4) (Musculoskeletal and connective tissue disorders) | 0 | 1
Dehydration (General disorders) | 1 | 0 — Grade 3
Febrile neutropenia, Diarrhea, Hand foot skin reaction, Acute renal failure (General disorders) | 1 | 0 — Grade 3
Pneumonia (Infections and infestations) | 1 | 0 — Grade 3
Ulcer gastric (Gastrointestinal disorders) | 1 | 0 — Grade 3
Hyperbilirrubinemia (Blood and lymphatic system disorders) | 1 | 0 — Grade 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xeloda (Capecitabine) (N=436) | Observation (N=425)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 0 — Grade 4
LYMPHOPENIA (Blood and lymphatic system disorders) | 3 | 1 — Grade 3
LYMPHOPENIA (Blood and lymphatic system disorders) | 19 | 6 — Grade 2
LYMPHOPENIA (Blood and lymphatic system disorders) | 40 | 26 — Grade 1
BILIRUBIN (Metabolism and nutrition disorders) | 1 | 0 — Grade 4
DIARRHEA (Gastrointestinal disorders) | 1 | 0 — Grade 4
DIARRHEA (Gastrointestinal disorders) | 14 | 0 — Grade 3
DIARRHEA (Gastrointestinal disorders) | 45 | 2 — Grade 2
DIARRHEA (Gastrointestinal disorders) | 94 | 4 — Grade 1
AST, SGOT (Metabolism and nutrition disorders) | 1 | 0 — Grade 4
AST, SGOT (Metabolism and nutrition disorders) | 8 | 0 — Grade 2
AST, SGOT (Metabolism and nutrition disorders) | 74 | 23 — Grade 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 — Grade 4
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 — Grade 3
URIC ACID, SERUM-HIGH (Metabolism and nutrition disorders) | 0 | 1 — Grade 4
URIC ACID, SERUM-HIGH (Metabolism and nutrition disorders) | 7 | 4 — Grade 1
IRREGULAR MENSES (Reproductive system and breast disorders) | 57 | 55 — Grade 3
IRREGULAR MENSES (Reproductive system and breast disorders) | 7 | 6 — Grade 2
IRREGULAR MENSES (Reproductive system and breast disorders) | 5 | 6 — Grade 1
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 82 | 0 — Grade 3
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 109 | 1 — Grade 2
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 115 | 2 — Grade 1
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 1 | 0 — Grade 3
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 54 | 12 — Grade 2
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 81 | 46 — Grade 1
NEUTROPHILS/GRANULOCYTES (Blood and lymphatic system disorders) | 8 | 0 — Grade 3
NEUTROPHILS/GRANULOCYTES (Blood and lymphatic system disorders) | 50 | 8 — Grade 2
NEUTROPHILS/GRANULOCYTES (Blood and lymphatic system disorders) | 67 | 38 — Grade 1
FATIGUE (General disorders) | 13 | 0 — Grade 3
FATIGUE (General disorders) | 48 | 10 — Grade 2
FATIGUE (General disorders) | 111 | 38 — Grade 1
HEMOGLOBIN (Blood and lymphatic system disorders) | 1 | 0 — Grade 3
HEMOGLOBIN (Blood and lymphatic system disorders) | 19 | 0 — Grade 2
HEMOGLOBIN (Blood and lymphatic system disorders) | 87 | 27 — Grade 1
NAUSEA (Gastrointestinal disorders) | 4 | 0 — Grade 3
NAUSEA (Gastrointestinal disorders) | 15 | 0 — Grade 2
NAUSEA (Gastrointestinal disorders) | 84 | 6 — Grade 1
ALT, SGPT (Metabolism and nutrition disorders) | 1 | 0 — Grade 3
ALT, SGPT (Metabolism and nutrition disorders) | 15 | 1 — Grade 2
ALT, SGPT (Metabolism and nutrition disorders) | 69 | 27 — Grade 1
NEUROPATHY: SENSORY (Nervous system disorders) | 3 | 1 — Grade 3
NEUROPATHY: SENSORY (Nervous system disorders) | 13 | 3 — Grade 2
NEUROPATHY: SENSORY (Nervous system disorders) | 50 | 21 — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2009-09-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT00130533/Prot_000.pdf
  • Statistical Analysis Plan (2010-05-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT00130533/SAP_001.pdf